CLINICAL TRIAL: NCT02063165
Title: Healthy Oils for Women: Reducing Visceral Adipose Tissue in Women with Metabolic Syndrome (HOW Study)
Brief Title: Healthy Oils for Women (HOW Study)
Acronym: HOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Corr-Jensen, LLC provided some of the study oil from Arista Industries, Inc (Unknown)
Responsible Party: Principal Investigator, Martha Belury, Carol S. Kennedy Professor of Nutrition, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012H0259; 2011-039 (Other Grant/Funding Number: Ohio Agricultural Research and Development Center)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome
Keywords: Safflower Oil; Linoleic Acid; Dyslipidemia; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Linoleic Acid (Experimental)
  Interventions: Dietary Supplement: High Linoleic Safflower Oil

INTERVENTIONS:
Dietary Supplement: High Linoleic Safflower Oil — 2 tsp per day (~10g of oil)

SUMMARY:
The purpose of this study is to understand the role of a dietary oil to alter chronic disease risk factors in women who are at risk for heart disease and/or diabetes. The investigator's previous study showed that safflower oil reduced trunk fat mass in women with diabetes. The investigators believe safflower oil can also attenuate criteria of metabolic syndrome through reduction in trunk fat mass.

DETAILED DESCRIPTION:
The long-term goal is to develop effective and novel dietary and lifestyle strategies to reduce the progression of metabolic syndrome to chronic diseases such as coronary heart disease. The rationale for conducting this research study is that there are few effective strategies that target changes in body composition and metabolism as a means to attenuate metabolic syndrome. The investigators plan to test the central hypothesis and accomplish the overall objective of this research by pursuing the following three specific aims.

Specific Aim 1: Quantify the extent that linoleic acid reduces trunk adipose mass in women with metabolic syndrome.

Specific Aim 2: Measure changes in visceral adipose tissue

Specific Aim 3: Determine the time-dependent effect of linoleic acid to increase adiponectin levels.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Post-menopausal (cessation of menses ≥12 months)
* Age ≥ 50 and ≤ 69 years
* At Least one of the following metabolic syndrome criteria

  * Elevated triglycerides (>150mg/dl)
  * Reduced HDL-C (<50mg/dl)
  * Elevated blood pressure (>130mm Hg systolic or > 85 mm Hg diastolic)
  * Elevated blood glucose (>100mg/dl and <126mg/dl)
* Obese (BMI ≥ 30 kg/m² and ≤ 55 kg/m²)

  * Stable medical therapy for past 3 months
* Stable body weight (within ± 2 kg) for past 3 months
* Waist circumference >88cm (35 inches)

Exclusion Criteria:

* Substance abuse
* Current/previous diagnosis of type 2 diabetes or fasting blood glucose ≥126 mg/dL
* Current use of medications or supplements known to affect body composition
* Current or previous use of oral hypoglycemic agents or exogenous insulin.
* Impaired cognitive function
* Current or previous diagnosis of renal, heart, or circulatory disease
* Gastrointestinal diseases or disorders

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in trunk adipose mass | Baseline and Week 16 (end of the study)

SECONDARY OUTCOMES:
Changes in Alpha and Gamma Tocopherol Levels | Baseline through Week 16 (end of the study)
Changes in mood | Baseline through Week 16 (end of the study)
  Mood questionnaires will be completed at each study visit
Changes in Lipid Profile | Baseline through Week 16 (end of the Study)
Oil Supplementation Compliance | Baseline through Week 16 (end of the study)
  Plasma and red blood cell fatty acid composition will be analyzed. Returned oil containers will be weighed to estimate oil consumption.
Changes in glycemic control | Baseline through Week 16 (end of the study)
  Serum glucose and insulin levels will be analyzed
Changes in lean mass | Baseline and Week 16 (end of the study)
Changes in visceral adipose tissue | Baseline and Week 16 (end of study)
Changes in adipocytokine levels | Baseline through Week 16 (end of the study)
  Adiponectin, leptin, and IL-6 will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Martha A Belury, PhD, RD, Principal Investigator — The Ohio State University, Department of Human Sciences, Human Nutrition Program
Locations (1):
- The Ohio State University Exercise Physiology Lab, Columbus, Ohio, United States

REFERENCES:
- [Derived] Cole RM, Puchala S, Ke JY, Abdel-Rasoul M, Harlow K, O'Donnell B, Bradley D, Andridge R, Borkowski K, Newman JW, Belury MA. Linoleic Acid-Rich Oil Supplementation Increases Total and High-Molecular-Weight Adiponectin and Alters Plasma Oxylipins in Postmenopausal Women with Metabolic Syndrome. Curr Dev Nutr. 2020 Aug 21;4(9):nzaa136. doi: 10.1093/cdn/nzaa136. eCollection 2020 Sep. PMID 32923921